CLINICAL TRIAL: NCT02817191
Title: Effects of Holy-Comod and Tears Naturale Forte on Ocular Surface and Tear Inflammatory Mediators in Patients After Phaco+IOL
Brief Title: Effects of Holy-Comod and Tears Naturale Forte in Patients After Phaco+IOL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xingwu Zhong, MD PhD, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-005
Record Dates: First submitted 2016-06-26; First posted 2016-06-29 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Age-related Cataract
Keywords: age-related cataract; Holy-Comod; Tears Naturale Forte; phacoemulsification; inflammatory mediators
MeSH Terms: interventions — Tobramycin; Dexamethasone; Tobramycin, Dexamethasone Drug Combination; methylacetylene

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hylo-Comod (Experimental): The patients used Hylo-Comod eye drop after phaco+IOL in this group.
  Interventions: Drug: Hylo-Comod eye drop
- Tears Naturale Forte (Experimental): The patients used Tears Naturale Forte eye drop after phaco+IOL in this group.
  Interventions: Drug: Tears Naturale Forte eye drop

INTERVENTIONS:
Drug: Hylo-Comod eye drop — The patients were administrated Hylo-Comod eye drop four times a day after Phaco+IOL
  Other Names: 0.3% tobramycin/dexamethasone (TobraDex, Alcon)
  Arms: Hylo-Comod
Drug: Tears Naturale Forte eye drop — The patients were administrated Tears Naturale Forte eye drop four times a day after Phaco+IOL
  Other Names: 0.3% tobramycin/dexamethasone (TobraDex, Alcon)
  Arms: Tears Naturale Forte

SUMMARY:
The purpose of the study it to compare the effects of Holy-Comod and Tears Naturale Forte on ocular surface and tear inflammatory mediators in patients after Phaco+IOL.

ELIGIBILITY:
Inclusion Criteria:

* 60-72 years old
* classification of lens nucleus is LOCS Ⅱ

Exclusion Criteria:

* patients with previous history of ocular surgery, corneal diseases,uveitis ,ocular hypertension or glaucoma ,systemic diseases.

Ages: 60 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
scale of Schirmer I test | up to 2 months after surgery
scale of corneal fluorescein staining | up to 2 months after surgery
scale of noninvasive tear breakup time | up to 2 months after surgery
questionnaire of ocular surface disease index | up to 2 months after surgery
scale of central corneal sensitivity | up to 2 months after surgery
scale of tear meniscus height | up to 2 months after surgery
concentration of Interleukin-1α | up to 2 months after surgery
concentration of tumor necrosis factor-α | up to 2 months after surgery
concentration of nerve growth factor | up to 2 months after surgery
concentration of interferon-γ | up to 2 months after surgery
concentration of transforming growth factor-β1 | up to 2 months after surgery
concentration of matrix metalloproteinase-9 | up to 2 months after surgery

SECONDARY OUTCOMES:
Correlation Between Inflammatory Mediators and Ocular Surface Changes | up to 2 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Xingwu Zhong, MD, PhD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Hainan Eye Hospital, Zhongshan Ophthalmic Center of Sun Yat-sen University, Haikou, Hainan, China